CLINICAL TRIAL: NCT06524414
Title: A Phase 2, Randomized, Double-Blind Trial to Evaluate the Safety, Tolerability, and Immunogenicity of a Multivalent Pneumococcal Conjugate Vaccine in Healthy Infants
Brief Title: A Study to Learn About How a New Pneumococcal Vaccine Works in Infants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4931002; NCT06524414 (Registry Identifier: ClinicalTrials.gov); 2025-000081-28 (EudraCT Number)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1 PG4 (Experimental): Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- Group 1 20-valent pneumococcal conjugate vaccine (20vPnC) (Active Comparator): 20-valent pneumococcal conjugate vaccine (20vPnC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC)
- Group 2 PG4 (Experimental): Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- Group 2 20-valent pneumococcal conjugate vaccine (20vPnC) (Active Comparator): 20-valent pneumococcal conjugate vaccine (20vPnC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC)
- Group 3 PG4 (Experimental): Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- Group 3 20-valent pneumococcal conjugate vaccine (20vPnC) (Active Comparator): 20-valent pneumococcal conjugate vaccine (20vPnC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC)
- Group 4 PG4 (Experimental): Multivalent Pneumococcal Vaccine
  Interventions: Biological: PG4
- Group 4 15-valent pneumococcal conjugate vaccine (PCV15) (Active Comparator): 15-valent pneumococcal conjugate vaccine (PCV15)
  Interventions: Biological: 15-valent pneumococcal conjugate vaccine (PCV15)

INTERVENTIONS:
Biological: PG4 — Multivalent pneumococcal conjugate vaccine
  Arms: Group 1 PG4; Group 2 PG4; Group 3 PG4; Group 4 PG4
Biological: 20-valent pneumococcal conjugate vaccine (20vPnC) — 20-valent pneumococcal conjugate vaccine
  Other Names: Prevnar 20
  Arms: Group 1 20-valent pneumococcal conjugate vaccine (20vPnC); Group 2 20-valent pneumococcal conjugate vaccine (20vPnC); Group 3 20-valent pneumococcal conjugate vaccine (20vPnC)
Biological: 15-valent pneumococcal conjugate vaccine (PCV15) — 15-valent pneumococcal conjugate vaccine
  Other Names: PCV15
  Arms: Group 4 15-valent pneumococcal conjugate vaccine (PCV15)

SUMMARY:
The purpose of this study is to learn about the safety of a new pneumococcal vaccine and how the new pneumococcal vaccine helps to fight against germs in infants when compared to the pneumococcal vaccines that are currently in use, 20vPnC (Prevnar 20®) or another licensed pneumococcal vaccine.

To ensure that the new vaccine (PG4) stays stable, it is placed in a liquid mixture of sterile water and other substances (a solution). This study will also test if there is a difference in the safety and immune effects of the new pneumococcal vaccine when it is one type of solution compared to when it is in a different type of solution.

The immune response is how the body's cells; tissues and organs work together to protect the body from infection. Blood samples will be used to measure the amount of antibodies produced after the vaccination. Antibodies are proteins that protect you when an unwanted germ enters the body. This will help understand how well the new pneumococcal vaccine works. This vaccine can possibly provide protection against pneumococcal disease. Pneumococcal disease includes a variety of infections caused by a specific germ, Streptococcus pneumoniae.

This study is seeking participants who are:

* male or female infants who are 2 months of age,
* infants born at 36 weeks (about 8 and a half months) of pregnancy or later; and,
* said to be healthy by the study doctor

There are four groups in this study. All participants will be assigned to one of the four groups. All study vaccines will be given as a single shot into the left thigh muscle. Participants in the three groups will have 3 blood samples collected during the 1 and a half years they are in the study.

The first 400 participants who enter the study will be assigned to either Group 1 or Group 2. Half the participants in Group 1 and half the participants in Group 2 will receive 4 doses at 2, 4, 6, and 12 to 15 months of age of PG4 mixed in the first solution. The other half of the participants in Groups 1 and 2 will receive 4 doses of 20vPnC (Prevnar 20®) at 2, 4, 6, and 12 to 15 months of age. The main difference between Groups 1 and 2 is that participants in Group 2 will have the first blood sample collected at an earlier time than those in Group 1.

Once 400 participants have been assigned to Groups 1 and 2 then 100 new participants will be assigned to Group 3. Half the participants in Group 3 will receive PG4 in the second solution at 2, 4, 6, and 12 to 15 months of age. The other half of the participants in Groups 3 will receive 4 doses of 20vPnC (Prevnar 20®) at 2, 4, 6, and 12 to 15 months of age.

Once the 100 participants have been assigned to Group 3 then 300 new participants will be assigned to Group 4. Half the participants in Group 4 will receive PG4 in the first solution at 2, 4, 6, and 12 to 15 months of age. The other half of the participants in Group 4 will receive 4 doses of a licensed pneumococcal comparator vaccine at 2, 4, 6, and 12 to 15 months of age.

Participants will take part in this study for about 16 to 19 months (about 1 and a half years). During this time, participants will have 6 study clinic visits and 1 to 2 phone calls. At these study clinic visits, parent(s) or legal guardian(s) will be asked if the participant experienced any side effects. A side effect is an unintentional or unexpected reaction to a vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at >36 weeks of gestation and 2 months of age at the time of consent.
* Healthy infants determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis).
* Major known congenital malformation or serious chronic disorder.
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 605 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions within 7 days after each dose | Day 7
  Prompted local reactions after each dose
Percentage of participants reporting systemic events within 7 days after each dose | Day 7
  Prompted systemic reactions after each dose
Percentage of participants reporting adverse events (AEs) | Dose 1 to 1 month after Dose 3
  AEs occurring from Dose 1 to 1 month after Dose 2
Percentage of participants reporting AEs | Dose 4 to 1 month after Dose 4
  AEs occurring from Dose 4 to 1 month after Dose 4
Percentage of participants reporting serious adverse events (SAEs) | Dose 1 to 6 months after Dose 4
  SAEs occurring from Dose 1 to 6 months after Dose 4

SECONDARY OUTCOMES:
Pneumococcal immunoglobulin G (IgG) geometric mean concentrations (GMCs) | 1 month after Dose 4
  Pneumococcal IgG GMCs 1 month after Dose 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (61):
- United States (54):
  - Northwest Arkansas Pediatric Clinic, Fayetteville, Arkansas
  - The Children's Clinic, Jonesboro, Arkansas
  - Los Ninos Children's Medical Clinic, La Puente, California
  - Stanford University Medical Center, Palo Alto, California
  - Los Ninos Children's Medical Clinic, West Covina, California
  - Velocity Clinical Research, Washington DC, Washington D.C., District of Columbia
  - Riveldi Biomedical Research and Associates - Miami, Miami Lakes, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - The Iowa Clinic, Ankeny, Iowa
  - Cotton O'Neil Pediatrics, Topeka, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - All Children Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - LSUHSC Clinical Trials Office, Shreveport, Louisiana
  - Louisiana State University Health Sciences Shreveport, Shreveport, Louisiana
  - Ochsner/LSU Health Ambulatory Care Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - UMB/CVD, Frederick, Maryland
  - Pediatric Associates of Fall River, Fall River, Massachusetts
  - Boeson Research GTF, Great Falls, Montana
  - OBGYN Associates, Great Falls, Montana
  - Boeson Research KAL, Kalispell, Montana
  - Heart and Hands Midwifery and Family Practice, Kalispell, Montana
  - POEM Healthcare, Kalispell, Montana
  - Blue Moose Pediatrics, Missoula, Montana
  - Boeson Research MSO, Missoula, Montana
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Child Health Care Associates, East Syracuse, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Durham Pediatrics at North Duke Street, Durham, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Ohio Pediatric Research Assn., Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Coastal Pediatric Research, Summerville, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Javara - Privia Medical Group North Texas - Dallas, Dallas, Texas
  - Oak Cliff Research Company, LLC, Dallas, Texas
  - PAS Research - McAllen, Edinburg, Texas
  - Mercury Clinical Research - Pediatric Associates, Houston, Texas
  - University of Texas Medical Branch, League City, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Alliance for Multispecialty Research, LLC, Kaysville, Utah
  - Tanner Clinic - Kaysville, Kaysville, Utah
  - Alliance for Multispecialty Research, LLC, Layton, Utah
  - Tanner Clinic, Layton, Utah
  - AMR Clinical, Murray, Utah
  - Alliance for Multispecialty Research, LLC, Provo, Utah
  - AMR Clinical, Roy, Utah
  - AMR Clinical, South Jordan, Utah
  - AMR Clinical, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
- Puerto Rico (7):
  - Clinical Research Puerto Rico, Guayama
  - Ponce Medical School Foundation Inc., Ponce
  - BRCR Global Puerto Rico, San Juan
  - Caribbean Medical Research Center, San Juan
  - University of Puerto Rico - Medical Sciences Campus, San Juan
  - The Hispanic Alliance for Clinical and Translational Research, San Juan
  - San Miguel Medical, Trujillo Alto

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4931002